CLINICAL TRIAL: NCT00011297
Title: Alcohol Research Center - Treatment and Implications
Brief Title: Comparing Gabapentin and Lorazepam for Treating Alcohol Withdrawal
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NIAAAMAL1076106
Record Dates: First submitted 2001-02-15; First posted 2001-02-19 (Estimated); Last update posted 2006-10-23 (Estimated); Status verified 2006-10

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Gabapentin; Lorazepam

INTERVENTIONS:
Drug: gabapentin (Neurontin)
Drug: lorazepam (Ativan)

SUMMARY:
This study will evaluate a safe and useful medication for outpatient detoxification that is as effective as benzodiazepines in the short-term, and more effective in the protracted withdrawal period. Gabapentin (Neurontin) will be compared to a standard benzodiazepine, lorazepam (Ativan), for its effectiveness in treating alcohol withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for alcohol dependence and uncomplicated alcohol withdrawal syndrome.
* Subjects must be medically stable (not likely to require hospitalization for medical complications within 10 days).
* Have a clinical withdrawal assessment prior to study.
* Must be medically acceptable for study treatment. Considerations include no past or present physical disorder that is likely to deteriorate during participation. No ECG abnormality which would likely worsen during participation and no clinical laboratory abnormality that would also suggest deterioration during treatment.
* Able to read, write, and speak English.
* Have a negative urine drug screen for benzodiazepines or other sedative hypnotics, opiates, and stimulates prior to entering the study.

Exclusion Criteria:

* Current diagnosis of any other substance dependence syndrome other than alcohol dependence (excluding nicotine and caffeine dependence).
* Use of pharmacological agents within the last 14 days that are known to lower the seizure threshold or augment or decrease the alcohol withdrawal syndrome.
* History of alcohol withdrawal seizures, epilepsy or delirium tremens.
* Diagnosis of schizophrenia, bipolar disorder or dementia.
* Liver function tests higher than normal.
* History of hepatic encephalopathy, jaundice, ascites, diabetes, or renal disease.
* Females who are pregnant or nursing.
* Subjects with known sensitivity of previous adverse reaction to gabapentin, lorazepam, or other benzodiazepines.
* History of severe GI disease which might render absorption of the medication difficult or produce medical instability of the patient during detoxification which would include active peptic ulcer disease, ulcerative colitis, regional colitis, or evidence by history or physical exam of GI bleeding.
* Unable to provide an informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Study Completion 2005-12

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States